CLINICAL TRIAL: NCT05768399
Title: The Role of Biomarkers in the Occurrence and Development of Asthma
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Fengxia Ding, Reseacher, Children's Hospital of Chongqing Medical University
Other Study IDs: File No.2023.225
Record Dates: First submitted 2023-02-07; First posted 2023-03-14 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Asthma in Children
Keywords: asthma; children; biomarkers
MeSH Terms: conditions — Asthma | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma group: Children with asthma diagnosed by a respiratory physician
  Interventions: Diagnostic Test: The level of biomarkers in Peripheral blood
- Control group: Children without respiratory disease or inflammatory diseases
  Interventions: Diagnostic Test: The level of biomarkers in Peripheral blood

INTERVENTIONS:
Diagnostic Test: The level of biomarkers in Peripheral blood — All participants will be extracted 5ml peripheral blood into the anticoagulant tube by nurses and the peripheral blood will be detected for biomarkers of asthma. Children with asthma will take pulmonary function, blood test and specific IgE test etc. The lung function test will be performed by professional technicians and the results will be interpreted by specialists. The blood test and specific IgE test will be collected by specialist nurses and the results will be issued by professional inspectors. Children with asthma and their guardians will be asked for filling the questionnaire of Childhood Asthma Control Test (C-ACT). And then the doctor will check and calculate the scores after completion.
  Other Names: pulmonary function, blood test, specific IgE

SUMMARY:
To study the expression level of biomarkers such as GITRL in peripheral blood of children with asthma and analyze their correlation with the severity of asthma. To study the predictive value of biomarkers level for the occurrence and development of asthma. And to provide supplementary detection means and predictive indicators for the diagnosis of asthma and the severity of asthma.

DETAILED DESCRIPTION:
Recruit 30 children with asthma and 30 healthy children based on the consent of the children and their parents or their guardian. Collect and record general information such as name, age, time of first diagnosis, allergens or triggers, daily dosage and frequency of asthma control drugs, home address and contact information. Collect 5 ml of blood sample for the detect of the biomarkers. Asthma severity was assessed using pulmonary function by spirometry and score of C-CAT. Finally study the correlation between the level of biomarkers and asthma severity and the role of biomarkers in the occurrence and development of asthma.

ELIGIBILITY:
Inclusion Criteria:

* In line with the diagnostic criteria in the Guidelines for the Diagnosis and Prevention of Bronchial Asthma in Children (2016 Edition)
* Age: 4-12 years old for new diagnosis or recurrent episodes
* Typical clinical manifestations and complete clinical data
* Family members or guardians of children with informed research and signed consent
* All healthy control subjects had no history of lung disease, allergic rhinitis or any other atopic disease

Exclusion Criteria:

* Suffering from other respiratory diseases (such as bronchiectasis, allergic rhinitis, respiratory failure, tuberculosis, obstructive airway disease) or other inflammatory diseases.
* Abnormal development of congenital airway and lung tissue
* History of immunosuppressant or glucocorticoid use in the first 4 weeks
* Suffering from other endocrine system and immune system diseases
* Incomplete clinical data or examinations.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with typical asthma symptoms, such as cough, wheezing, chest tightness, dyspnea and abnormal lung function tests, were diagnosed with asthma by a respiratory doctor
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The level of biomarkers | 2years
  All participants will be extracted 5ml peripheral blood into the anticoagulant tube by nurses and the peripheral blood will be detected for biomarkers of asthma using RT-qPCR、 ELISA、 Flow cytometry and other methods.

SECONDARY OUTCOMES:
Pulmonary function（FEV1%） | 2 years
  The correlation of pulmonary function （FEV1） and the level of biomarkers in children with asthma.The lung function test will be performed by professional technicians and the results will be interpreted by specialists.
Pulmonary function（FVC%） | 2 years
  The correlation of pulmonary function （FVC%） and the level of biomarkers in children with asthma.The lung function test will be performed by professional technicians and the results will be interpreted by specialists.
Pulmonary function（FEV1/FVC） | 2 years
  The correlation of pulmonary function （FEV1/FVC） and the level of biomarkers in children with asthma.The lung function test will be performed by professional technicians and the results will be interpreted by specialists.
Pulmonary function（PEF%） | 2 years
  The correlation of pulmonary function （PEF%） and the level of biomarkers in children with asthma.The lung function test will be performed by professional technicians and the results will be interpreted by specialists.
specific IgE | 2 years
  The correlation of blood specific IgE and the level of biomarkers in children with asthma
Peripheral blood eosinophil count | 2 years
  The correlation of peripheral blood eosinophil count and the level of biomarkers in children with asthma
Childhood Asthma Control Test (C-ACT) | 2 years
  The correlation of the score of C-ACT and the level of biomarkers in children with asthma. Children with asthma and their guardians will be asked for filling the questionnaire of Childhood Asthma Control Test (C-ACT). And then the doctor will check and calculate the scores after completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoqing Zhang, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No